CLINICAL TRIAL: NCT07145255
Title: A Multicenter, Open-label Phase 1/2 Dose Finding, Safety, and Pharmacokinetic Study of MBRC-201, an Antibody-drug Conjugate, in Advanced Refractory Solid Tumors
Brief Title: Phase 1/2 Dose Finding, Safety and PK Study in Advanced Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MBrace Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBRC-201-001
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Castration-resistant Prostate Cancer; Breast Cancer; Colo-rectal Cancer; Lung Cancer (Non-Small Cell); Pancreas Cancer, Duct Cell Adenocarcinoma
Keywords: ADC; prostate cancer; breast cancer; colorectal cancer; non-small cell lung cancer; MBrace
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a (Experimental): Dose Escalation
  Interventions: Drug: ADC
- Phase 1b (Experimental): Dose Expansion
  Interventions: Drug: ADC
- Phase 2 (Experimental): Recommended Phase 2 Dose
  Interventions: Drug: ADC

INTERVENTIONS:
Drug: ADC — MBRC-201 ADC

SUMMARY:
This is a multicenter, open-label FIH, Phase 1a (dose escalation), Phase 1b (dose expansion) and Phase 2 study in patients with advanced metastatic solid tumors refractory to standard treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label FIH, Phase 1a (dose escalation), Phase 1b (dose expansion) and Phase 2 study in patients with advanced metastatic solid tumors refractory to standard treatment.

Phase 1a will characterize safety and identify potential optimal biologically relevant doses (OBRDs), Recommended Phase 2 Doses (RP2Ds), and the maximum tolerated dose (MTD) of MBRC-201 at one or more dosing regimens.

Phase 1b will evaluate the safety and preliminary clinical activity of MBRC-201 at the potential OBRDs, RP2Ds, and dosing regimens identified in Phase 1a. The initial Phase 2 portion will begin when the RP2D has been determined from Phase 1a and Phase1b data. Phase 1b will enroll at least 4 expansion cohorts of approximately 20 patients per cohort (n ≈ 80 total) with the following tumor types: patients with mCRPC with confirmed adenocarcinoma histology, patients with advanced metastatic NSCLC refractory to standard treatment, patients with advanced metastatic breast cancer (TNBC, HR+/HER2-low or -negative, or HR-/HER2-low) refractory to standard treatment, and patients with advanced metastatic CRC or PDAC refractory to standard treatment.

The initial Phase 2 will enroll approximately 30 patients to further evaluate antitumor activity and safety of MBRC-201 at the RP2D determined during Phase 1b. Phase 2 will enroll patients in tumor-specific cohorts from the indications evaluated in Phase 1a/1b.

Phase 1a, Phase 1b and Phase 2 will characterize single and multiple-dose PK profiles and evaluate incidence and persistence of anti-MBRC-201 antibody (Ab) [ADA] formation. Safety will be assessed at each dose escalation in Phase 1a and ad hoc throughout Phase 1b and Phase 2.

A Safety Review Committee (SRC), consisting of the site investigators and representatives from the Sponsor will monitor patient safety and make dosing recommendations throughout the study.

The duration of the study (e.g., from the first patient enrolled through completion of LTFU data collection) is estimated to be approximately 48 months. There will also be long-term follow-up (LTFU) for safety, disease status, and survival assessments, which will continue until death or lost to follow-up, withdrawal of consent for further follow-up, or study termination whichever occurs first

ELIGIBILITY:
Inclusion Criteria: Patients are eligible to be included in the study only if all of the following criteria apply:

1. Provide written consent on an informed consent form (ICF), approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific evaluation. Patients should have the ability to read and understand the ICF, ask for any clarifications from the study staff, and be able to comply with all planned study procedures.
2. 18 years of age or older at the time of informed consent.
3. Female patients must be at least 2 years postmenopausal (defined as 2 years without menses), surgically sterile (at least 6 months prior to dosing; must be documented) or patients of childbearing potential under the following conditions:

   * Must be nonlactating and have a negative serum (preferred) or urine pregnancy test results within 72 hours prior to the first dose of MBRC-201.
   * Must agree not to try to become pregnant during the study and for at least 6 months after the final dose of MBRC-201
   * Must agree to practice effective contraception (must agree to use 2 forms of contraception, 1 of which must be a barrier method) and willing to continue to use effective contraception for the duration of study participation and for 6 months after the final dose of study drug.
4. Male patients whose partners are of childbearing potential must agree to use effective contraception (must agree to use 2 forms of contraception, 1 of which must be a barrier method) (Section 10.4) for the duration of study participation and for 6 months after the final dose of study drug.
5. Have a histologic or cytologic diagnosis of malignant solid tumor for which there are no standard-of-care treatment options known to confer a clinical benefit or for which the patient is ineligible or declines (except for Phase 1b-Cohort A).

   A. For Phase 1a dose escalation: Patients must have one of the following tumor types:

   i. mCRPC, breast cancer (TNBC, HR+/HER2-negative or HER2-low, HR-/HER2+), CRC, NSCLC, or PDAC

   B. For Phase 1b: Patients must have one of the following tumor types:

   i. Cohort A: Histologic or cytologic diagnosis of mCRPC (with confirmed adenocarcinoma histology) refractory to standard treatment.

   Patients must have had prior exposure to at least one novel AR-targeted therapy (e.g., abiraterone acetate, enzalutamide, apalutamide, darolutamide). Prior taxane or lutetium Lu 177 vipivotide tetraxetan is acceptable but not required.

   ii. Cohort B: Histologic or cytologic diagnosis of advanced metastatic NSCLC refractory to standard treatment.

   iii. Cohort C: Histologic or cytologic diagnosis of advanced metastatic breast cancer (TNBC, HR+/HER2-negative or HER2-low, HR-/HER2+) refractory to standard treatment.

   iv. Cohort D: Histologic or cytologic diagnosis of advanced metastatic CRC, PDAC refractory to standard treatment. The Sponsor may add or remove specific tumor indications based on emerging, real-time study results.
6. Availability of a tumor tissue sample (formalin-fixed paraffin-embedded [FFPE]) must be confirmed if feasible. Patients without tumor sample may be eligible with medical monitor approval. Tumor biopsies are not required and should not be performed to assess eligibility.
7. For Dose Escalation (Phase 1a), patients may have evaluable disease or measurable disease according to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1. For both Dose Expansion (Phase 1b) and Phase 2, patients must have measurable disease according to RECIST v1.1
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
9. Life expectancy ≥ 3 months
10. Patient must have adequate organ and marrow function as defined below.

    * Absolute neutrophil count (ANC) ≥ 1500/uL
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Platelet count ≥ 100,000/uL
    * International normalized ratio (INR) < 1.5 (or ≤ 3.0 if on therapeutic anticoagulation)
    * Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min by the CKD-EPI or similar equation or as measured by 24-hour urine collection
    * Total bilirubin ≤ 1.5 × ULN [or ≤ 3-times ULN for patients with Gilbert's disease or documented hepatic tumor involvement]
    * ALT and AST ≤ 3 × ULN [or ≤ 5-times ULN for patients with documented hepatic tumor involvement]

Exclusion Criteria: Patients are excluded from the study if any of the following criteria apply:

1. History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Allowed exceptions are patients with:

   1. Non-melanoma skin cancer considered completely cured;
   2. Localized prostate cancer treated with curative intent with no evidence of progression;
   3. Low-risk or very low-risk (per standard clinical guidelines) localized prostate cancer under active surveillance without immediate intent to treat;
   4. Malignancy that is otherwise considered cured with minimal risk of recurrence.
2. Known or suspected sensitivity to any of the ingredients of the investigational product MBRC-201.
3. Active cerebral/meningeal disease related to the underlying malignancy. Patients with a history of cerebral/meningeal disease related to the underlying malignancy are allowed if prior central nervous system disease has been treated and the patient is clinically stable. (defined as not having received steroid treatment for symptoms related to cerebral/meningeal disease for at least 2 weeks prior to the first dose of study drug and with no ongoing related AEs).
4. Any uncontrolled viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study drug, unless deemed not clinically significant by the investigator (e.g., onychomycosis). Routine antimicrobial prophylaxis is permitted.
5. Active or symptomatic viral hepatitis, including patients with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months). Patients who have been treated for hepatitis C infection or who have spontaneously recovered are permitted.
6. Patients with HIV infection with 1 or more of the following:

   * Acquired immunodeficiency syndrome (AIDs)-defining opportunistic infection within 6 months of the start of screening
   * A change in antiretroviral therapy within 3 months of the start of screening and viral load > 500 copies/mL
   * Receiving antiretroviral therapy that may interfere with study drug
   * CD4 count < 350 at screening
7. Thromboembolic events and/or bleeding disorders ≤ 14 days (e.g., venous thromboembolism [VTE] or pulmonary embolism [or PE]) prior to the first dose of study drug
8. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study drug
9. A baseline QT (time from the beginning of the Q wave to the end of the T wave) interval as corrected by Fridericia's formula (QTcF) > 470 msec or patients with risk factors for Torsades de pointes
10. Uncontrolled Inflammatory Bowel Disease (IBD)
11. A history of (non-infectious) ILD/pneumonitis requiring steroid therapy, or active ILD/pneumonitis, or clinically suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
12. Uncontrolled autoimmune disease or syndrome
13. Active ocular surface disease at screening, including confluent superficial keratitis, cornea epithelial defect, corneal ulcer or stromal opacity or any components of the ophthalmologic history which, in the investigator's opinion, may place the patient at significant risk. Cataracts alone are not an exclusion criterion.
14. Any anticancer therapy within 14 days prior to the first dose of study drug, including: small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy, radiotherapy, or any other agents to treat cancer (anti-hormonal therapy given for advanced prostate cancer or as adjuvant therapy for early stage, HR positive breast cancer is not considered cancer therapy for the purpose of this protocol).
15. Use of any investigational drug within 14 days prior to the first dose of study drug.
16. For Phase 1b and Phase 2: prior treatment with an ADC with a camptothecin (CPT) payload, such as Enhertu (trastuzumab deruxtecan), Datroway (datopotamab deruxtecan), or Trodelvy (sacituzumab govitecan). Prior treatment with irinotecan and other non-ADC topoisomerase inhibitors is allowed in all phases of the study.
17. Current use of any prohibited concomitant medication(s).
18. Major surgery within 28 days prior to first dose of study drug.
19. Patients who have not recovered from AEs due to prior anticancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia
20. Any medical, psychiatric, addictive, or other kind of disorder which compromises the ability of the patient to give written informed consent and/or to comply with procedures.
21. Condition or situation which, based on Investigator or Sponsor assessment, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study.
22. Other serious underlying medical condition that would impair the patient's ability to receive or tolerate the planned treatment and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of adverse events (AEs) | From Enrollment through treatment and long term follow-up (approximately 24 months)
  • TEAEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.0.
• Incidence and prevalence of Dose-limiting Toxicities (DLTs) and cumulative safety by dose level | 21 days
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, hematologic toxicity, and Non-hematologic (laboratory) toxicities
Duration of Response (DOR) | Approximately 24 months
  will be defined as the time from the first documentation of an objective tumor response (CR or PR) to the first documentation of tumor progression or to death due to any cause, whichever comes first, whichever comes first as defined by RECIST version 1.1.
Disease Control Rate (DCR) | Approximately 24 months
  DCR will be defined as the proportion of patients with best overall response of CR, PR, or stable disease (SD), whichever comes first as defined by RECIST version 1.1.
Progression Free Survival (PFS) | Approximately 24 months
  PFS will be defined as the time from the start of any study treatment to first documentation of disease progression or to death due to any cause, whichever comes first as defined by RECIST version 1.1.

SECONDARY OUTCOMES:
To evaluate the antitumor activity of MBRC-201 at the RP2D | Approximately 24 months
  Investigator-assessed ORR by RECIST v1.1
To evaluate preliminary antitumor activity of MBRC-201 at potential RP2D, OBRDs, and dosing regimens | approximately 24 months
  Investigator-assessed ORR by Response Evaluation Criteria in Solid Tumor (RECIST) v1.1

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - START, Midwest, Grand Rapids, Michigan
  - START, Astera, East Brunswick, New Jersey
  - NEXT, Dallas, Irving, Texas
  - START San Antonio, San Antonio, Texas
  - START, Mountain Region, West Valley City, Utah
  - NEXT, Virginia, Fairfax, Virginia